CLINICAL TRIAL: NCT00006250
Title: Randomized Trial of MCD Versus FMD in Untreated Advanced Follicular Lymphoma
Brief Title: Combination Chemotherapy in Treating Patients With Newly Diagnosed Stage III or Stage IV Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lymphoma Trials Office (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068182; BNLI-MCD/FMD; EU-20035
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2007-03

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Chlorambucil; Dexamethasone; fludarabine phosphate; Mitoxantrone

INTERVENTIONS:
Drug: chlorambucil
Drug: dexamethasone
Drug: fludarabine phosphate
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. It is not yet known which combination chemotherapy regimen is more effective for non-Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different combination chemotherapy regimens in treating patients who have stage III or stage IV non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival rate, progression free survival rate, clinical and molecular remission rates, and time to treatment failure in patients with newly diagnosed stage III or IV follicular non-Hodgkin's lymphoma treated with chlorambucil, mitoxantrone, and dexamethasone versus fludarabine, mitoxantrone, and dexamethasone.
* Compare the efficacy and tolerability of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to International Prognostic Index score [low risk (score 1) vs intermediate low risk (score 2) vs intermediate high risk (score 3) vs high risk (score 4 or 5)]. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive mitoxantrone IV on day 1, oral chlorambucil on days 1-10, and oral dexamethasone on days 1-5.
* Arm II: Patients receive mitoxantrone and dexamethasone as in arm I and fludarabine IV on days 1-3.

Treatment continues every 4 weeks for 4-8 courses.

Patients are followed at 3, 6, and 12 months, every 6 months for 1 year, and then annually thereafter until clinical relapse.

PROJECTED ACCRUAL: A total of 500 patients (250 per arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven newly diagnosed stage III or IV follicular non-Hodgkin's lymphoma

  * REAL classification grade I, II, or III
* Treatment necessity indicated by presence of the following:

  * B symptoms
  * Bone marrow failure
  * Bulky or progressive disease
  * Compression syndromes
* No CNS involvement

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* No autoimmune hemolytic anemia or active hemolysis
* Direct Coombs' negative

Hepatic:

* Alkaline phosphatase no greater than 2.5 times upper limit of normal (ULN)*
* Bilirubin no greater than 2.5 times ULN* NOTE: *Unless attributable to lymphoma

Renal:

* Creatinine no greater than 2.5 times ULN (unless attributable to lymphoma)

Cardiovascular:

* No severe cardiac failure
* Ejection fraction at least 45%

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for at least 6 months after study
* HIV negative
* No prior malignancy except carcinoma in situ of the cervix or squamous cell skin cancer
* No other serious medical disease that would limit lifespan or ability to tolerate chemotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent systemic corticosteroids

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2000-05

PRIMARY OUTCOMES:
Time to treatment failure
Progression-free survival rate
Overall survival rate

SECONDARY OUTCOMES:
Clinical remission rate
Molecular remission rate

CONTACTS AND LOCATIONS:
Overall Officials: Andy Haynes, MD, Study Chair — Nottingham City Hospital
Locations (59):
- United Kingdom (59):
  - Stoke Mandeville Hospital, Aylesbury-Buckinghamshire, England
  - Basildon University Hospital, Basildon, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Bradford Hospitals NHS Trust, Bradford, England
  - Kent and Canterbury Hospital, Canterbury, England
  - St Helier Hospital, Carshalton, England
  - Saint Richards Hospital, Chichester, England
  - Walsgrave Hospital, Coventry, England
  - Dartford & Gravesham NHS Trust, Joyce Green Hospital, Dartford Kent, England
  - Derbyshire Royal Infirmary, Derby, England
  - Doncaster Royal Infirmary, Doncaster, England
  - Russells Hall Hospital, Dudley, England
  - Epsom General Hospital, Epsom Surrey, England
  - Northwick Park Hospital, Harrow, England
  - Wycombe General Hospital, High Wycombe, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Hull Royal Infirmary, Hull, England
  - Ipswich Hospital NHS Trust, Ipswich, England
  - West Middlesex University Hospital, Isleworth, England
  - Kettering General Hosptial, Kettering, Northants, England
  - Queen Elizabeth Hospital, Kings Lynn, England
  - Clinical Trials and Research Unit of the University of Leeds, Leeds, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Aintree University Hospital, Liverpool, England
  - St. Thomas' Hospital, London, England
  - St. Georges, University of London, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - University College of London Hospitals, London, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Derriford Hospital, Plymouth, England
  - Pontefract General Infirmary, Pontefract West Yorkshire, England
  - Oldchurch Hospital, Romford, England
  - Rotherham District General Hospital - NHS Trust, Rotherham, England
  - Pembury Hospital, Royal Tunbridge Wells, Kent, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Royal Hallamshire Hospital, Sheffield, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Staffordshire General Hospital, Stafford, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Taunton and Somerset Hospital, Taunton Somerset, England
  - Torbay Hospital, Torquay Devon, England
  - Hillingdon Hospital, Uxbridge, England
  - Sandwell General Hospital, West Bromwich, England
  - Good Hope Hospital Trust, West Midlands, England
  - New Cross Hospital, Wolverhampton, England
  - Worthing Hospital, Worthing, England
  - Yeovil District Hospital, Yeovil - Somerset, England
  - Cancer Care Centre at York Hospital, York, England
  - Centre for Cancer Research and Cell Biology at Belfast City Hospital, Belfast, Northern Ireland
  - Craigavon Area Hospital, Craigavon, Northern Ireland
  - Ulster Hospital, Dundonald, Northern Ireland
  - Pinderfields Hospital NHS Trust, Wakefield, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - University Hospital of Wales, Cardiff, Wales
  - Glan Clywd District General Hospital, Rhyl, Denbighshire, Wales
  - Singleton Hospital of the Swansea NHS Trust, Swansea, Wales